CLINICAL TRIAL: NCT07340333
Title: Reference Values and Hemodynamic Associations of Total Arterial Impedance Derived From PRAM Monitoring During Hemodynamically Stable Intraoperative Periods
Brief Title: Physiological Reference Values of Total Arterial Impedance Derived From PRAM Monitoring
Acronym: PRAM-ZTOT
Status: Completed | Type: Observational
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mehmet Akif Yilmaz, Principal Investigator, Ataturk University
Other Study IDs: ATAUNI-PRAM-ZTOT-2026; 2026/1 (Other: Atatürk University Clinical Research Ethics Committee)
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Intraoperative Hemodynamics
Keywords: Total arterial impedance; PRAM monitoring; Arterial load; Advanced hemodynamic monitoring; Pressure waveform analysis; Physiological reference values; Intraoperative hemodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Intraoperative PRAM Monitoring Cohort: Adult surgical patients with invasive arterial monitoring whose intraoperative hemodynamic data were retrospectively analyzed during predefined hemodynamically stable periods using PRAM-based waveform analysis.

SUMMARY:
Total arterial impedance (Ztot) is an advanced hemodynamic parameter that reflects the global arterial load opposing ventricular ejection by integrating both steady and pulsatile components of the arterial system. Although Ztot can be continuously derived from Pressure Recording Analytical Method (PRAM)-based monitoring, physiological reference values under stable clinical conditions are not well established.

This observational study aims to define patient-level physiological reference values for Ztot using intraoperative hemodynamic data obtained from PRAM-based arterial waveform analysis during hemodynamically stable periods. In addition, the study evaluates the associations between Ztot and key hemodynamic variables reflecting arterial load and cardiovascular performance.

High-resolution intraoperative data routinely recorded during standard clinical care are retrospectively analyzed. The findings of this study are intended to improve the interpretability of Ztot in advanced hemodynamic monitoring and to support future clinical and research applications.

DETAILED DESCRIPTION:
Total arterial impedance (Ztot) is a comprehensive descriptor of arterial load that integrates resistive, compliant, and pulsatile components of the arterial system. Unlike conventional pressure-based parameters, Ztot provides a more physiologically meaningful representation of the opposition encountered by ventricular ejection. Although Ztot can be continuously estimated using Pressure Recording Analytical Method (PRAM)-based arterial waveform analysis, standardized physiological reference values applicable to routine clinical practice are lacking.

This single-center, observational study is designed to establish patient-level reference values for PRAM-derived Ztot during hemodynamically stable intraoperative periods. The study retrospectively analyzes high-resolution intraoperative hemodynamic data obtained during routine clinical care. Adult surgical patients monitored with an invasive arterial catheter and PRAM-based hemodynamic monitoring are included in the analysis.

Hemodynamic stability is defined according to predefined physiological criteria, including ranges of mean arterial pressure, cardiac index, heart rate, stroke volume variation, cardiac cycle efficiency, and arterial waveform quality indicators. Only measurements meeting all stability criteria are considered eligible for analysis.

To account for repeated measurements within individuals, patient-level median values are used for all primary analyses. The physiological reference interval for Ztot is estimated using a non-parametric percentile-based approach. In addition, associations between Ztot and key hemodynamic variables related to arterial load and cardiovascular performance are explored using correlation analyses.

This study does not involve any interventions, treatment assignments, or changes to standard clinical management. The primary objective is descriptive and physiological, aiming to provide a reference framework that may enhance the clinical interpretability of Ztot in advanced hemodynamic monitoring. The results are expected to support future prospective and outcome-oriented research evaluating the role of Ztot in perioperative and critical care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) who underwent surgery with invasive arterial catheterization.
* Availability of intraoperative hemodynamic data recorded using PRAM-based arterial waveform monitoring.
* Presence of predefined hemodynamically stable intraoperative periods meeting physiological stability criteria.
* Adequate arterial waveform signal quality for PRAM-derived parameter analysis.

Exclusion Criteria:

* Age <18 years.
* Inadequate arterial waveform signal quality or missing PRAM-derived data.
* Absence of intraoperative periods fulfilling predefined hemodynamic stability criteria.
* Incomplete or corrupted intraoperative monitoring records.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult surgical patients who underwent routine intraoperative invasive arterial monitoring, from whom PRAM-based hemodynamic data were retrospectively analyzed during predefined hemodynamically stable intraoperative periods.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2026-01-30 (Actual); Primary Completion 2026-02-02 (Actual); Study Completion 2026-02-02 (Actual)

PRIMARY OUTCOMES:
Physiological reference interval of total arterial impedance (Ztot) | Intraoperative period
  Patient-level physiological reference interval (2.5th-97.5th percentiles) of PRAM-derived total arterial impedance (Ztot) calculated from intraoperative hemodynamic measurements obtained during predefined hemodynamically stable periods.

SECONDARY OUTCOMES:
Association between total arterial impedance and arterial load-related hemodynamic variables | Intraoperative period
  Correlation between patient-level total arterial impedance (Ztot) and arterial load-related hemodynamic variables, including effective arterial elastance and systemic vascular resistance.
Association between total arterial impedance and cardiovascular performance indices | Intraoperative period
  Association between patient-level total arterial impedance (Ztot) and indices of cardiovascular performance, including cardiac output, stroke volume, cardiac power output, and cardiac cycle efficiency.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional and ethical restrictions related to patient privacy and the retrospective nature of the study. The analyzed data consist of anonymized intraoperative monitoring records collected during routine clinical care. Aggregated and summary-level results are reported in publications, and additional information may be made available upon reasonable request and with appropriate institutional approval.

REFERENCES:
- [Background] Vlachopoulos C, O'Rourke M, Nichols WW. McDonald's Blood Flow in Arteries: Theoretical, Experimental and Clinical Principles. 6 ed. Boca Raton, FL: CRC Press; 2011.
- [Background] Kelly RP, Ting CT, Yang TM, Liu CP, Maughan WL, Chang MS, Kass DA. Effective arterial elastance as index of arterial vascular load in humans. Circulation. 1992 Aug;86(2):513-21. doi: 10.1161/01.cir.86.2.513. PMID 1638719
- [Background] Kass DA. Ventricular arterial stiffening: integrating the pathophysiology. Hypertension. 2005 Jul;46(1):185-93. doi: 10.1161/01.HYP.0000168053.34306.d4. Epub 2005 May 23. PMID 15911741
- [Background] Sunagawa K, Sagawa K, Maughan WL. Ventricular interaction with the loading system. Ann Biomed Eng. 1984;12(2):163-89. doi: 10.1007/BF02584229. PMID 6507965
- [Background] Westerhof N, Lankhaar JW, Westerhof BE. The arterial Windkessel. Med Biol Eng Comput. 2009 Feb;47(2):131-41. doi: 10.1007/s11517-008-0359-2. Epub 2008 Jun 10. PMID 18543011
- [Background] O'Rourke M, Adji A, Nichols WW, Vlachopoulos C, Edelman ER. Application of Arterial Hemodynamics to Clinical Practice: A Testament to Medical Science in London. Artery Res. 2017 Jun;18:81-86. doi: 10.1016/j.artres.2017.03.003. No abstract available. PMID 29861794
- [Background] de Keijzer IN, Scheeren TWL. Perioperative Hemodynamic Monitoring: An Overview of Current Methods. Anesthesiol Clin. 2021 Sep;39(3):441-456. doi: 10.1016/j.anclin.2021.03.007. Epub 2021 Jul 12. PMID 34392878
- [Background] Pinsky MR. Functional hemodynamic monitoring. Crit Care Clin. 2015 Jan;31(1):89-111. doi: 10.1016/j.ccc.2014.08.005. PMID 25435480